CLINICAL TRIAL: NCT06891079
Title: Videodensitometric Angiographic Assessment of AR in the Cath-lab for Intraprocedural Guidance of TAVI in CHINA-A Prospective, Randomized, Controlled, Open-label, Multi-centre, Non-inferiority Trial
Brief Title: Videodensitometric Angiographic Assessment of AR in the Cath-lab for Intraprocedural Guidance of TAVI in CHINA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OVAL GUIDE CHINA
Record Dates: First submitted 2025-02-16; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; transcatheter aortic valve implantation; videodensitometry; Paravalvular regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): TAVI procedure guided by post-implantation aortographic quantitative videodensitometric assessment.
  Interventions: Diagnostic Test: Videodensitometric guided
- Control arm (Active Comparator): TAVI procedure guided by post-implantation standard of care according to local practice.
  Interventions: Diagnostic Test: Stand of care guided

INTERVENTIONS:
Diagnostic Test: Videodensitometric guided — In the experimental arm, a TAVI device is implanted according to the local practice. Immediately after implantation, aortography is performed to quantitatively assess the aortic regurgitation (qAR). The aortography is analyzed using CAAS A-Valve (Pie-Medical, Maastricht, The Netherlands).
  •If qAR is >17%, we recommend that corrective post-TAVI manoeuvres (post-dilatation, valve-in-valve, etc.) will be performed and angiography is repeated for the assessment of aortic regurgitation. If the qAR ≤17%, whether corrective post-TAVI manoeuvres (post-dilatation, valve-in-valve, etc.) will be performed is left to the discretion of the operators. Inform operators of the results of qAR and the threshold criteria. Continuous qAR was stratified into categorical variables according to the following pre-determined threshold criteria: (1) none or trace (qAR <6%); (2) mild (6% to ≤17%); and (3) moderate or severe (>17%).
  At discharge, all the patients will undergo Cardiac magnetic resonance, the Car
  Arms: Experimental arm
Diagnostic Test: Stand of care guided — In the control arm, a TAVI device is implanted according to local practice. Immediately after implantation, TEE/TTE or aortography is performed as a part of usual practice.
  * The requirement of post-dilatation or any additional procedure is left to the discretion of the operator.
  * The operator judges the sufficient procedural outcome to end the procedure according to local practice.
  At discharge, all the patients will undergo Cardiac magnetic resonance, the Cardiac magnetic resonance-derived regurgitation fraction (CMR-RF) will be analyzed as the primary endpoint.
  Arms: Control arm

SUMMARY:
This clinical trial, a prospective, randomized, multicenter study, assigns patients to either videodensitometry-guided TAVI or conventional TTE/TEE-guided TAVI (stand of care), with the primary endpoint being regurgitation fraction measured by cardiac magnetic resonance (CMR) at discharge. Current AR assessment methods, like subjective visual grading or intraprocedural TTE, face limitations in objectivity and practicality, whereas videodensitometry offers real-time, quantitative feedback to guide corrective actions (e.g., post-dilation) during TAVI. If proven non-inferior, this approach could streamline workflows by reducing reliance on general anesthesia and complex imaging, potentially lowering complications and expanding accessibility, particularly in centers lacking advanced echocardiography resources.

DETAILED DESCRIPTION:
As the transcatheter aortic valve implantation (TAVI) procedure matures, complications such as paravalvular regurgitation (PVR), stroke, conduction disturbances, vascular complications, and annular rupture have been targeted for further improving the long-term outcome of TAVI. Paravalvular regurgitation (PVR) is associated with mortality following TAVI, even in those with mild PVR. Accurate procedural assessment of AR-critical for successful TAVI. Aortic root angiography, typically using Seller's visual grading, is the first screening tool used in most laboratories for the detection of post-implantation AR and guidance of timely corrective measures (e.g. post-dilation, valve-in-valve and, most recently, retrieval and reposition of the valve). However, the Sellers classification of aortic regurgitation (AR) is subjective. Some centers use transthoracic echo to confirm residual AR. However, performing transthoracic echo in the Cath-lab in a prone position is challenging. Previous studies have demonstrated that TAVI performed exclusively under angiographic guidance with backup TTE is feasible and associated with reasonably good outcomes, similar to those of angiography and TEE-guided procedures. Quantitative aortographic assessment of AR is important for procedural TAVI guidance to facilitate timely decision-making to avert AR using balloon post-dilatation, retrieval-reposition, or valve-in-valve implantation.

CAAS A-Valve (quantitative assessment of regurgitation with videodensitometry in the left ventricle outflow tract) is a new tool to quantify AR developed by Pie Medical. This tool is an angiographic methodology that proved to be accurate, feasible, reproducible, and predictive of outcomes after TAVI. After extensive validation of this new technology in two different cohorts (from the Brazilian TAVI registry and Bad-Segeberg, Germany), hereby we propose to apply this currently off-line technology to guide decision making in the Cath-lab during TAVI.

The present trial is a prospective, randomized, controlled, open-label, multi-center, non-inferiority trial. The primary objective of this trial is to determine whether TAVI procedure guided by videodensitometric assessment of aortography is non-inferior to TAVI implantation guided by Standard of care (usual practice) in terms of postprocedural quantitative aortic regurgitation. The primary endpoint of the study will be the Cardiac magnetic resonance-derived regurgitation fraction at discharge. This project is the first study to investigate the clinical utility of using video-densitometry in a randomized, controlled clinical trial to guide TAVI procedure. In centers with no current CAAS-A Valve software, Pie Medical will provide a research lease during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has aortic stenosis with indication of TAVI implantation as determined by Heart Team.
2. Patient is at least 18 years of age.
3. Signed informed consent. The patient understands and accepts clinical follow-up.

Exclusion Criteria:

1. Subject is not willing to provide an informed consent form, or whose legal heirs object to their participation in the study.
2. If the patient is not suitable for participating in the study, based on the evaluation by the operators.
3. Cardiogenic shock.
4. Significant comorbidities precluding clinical follow-up (as judged by investigators).
5. History of TAVI or SAVR.
6. Renal insufficiency (GFR/MDRD <45 ml/min), which precludes in operator's opinion contrast injection during repeat aortography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CMR-derived regurgitation fraction | at discharge 1 day, an average of 7days
  The Cardiac magnetic resonance-derived regurgitation fraction at discharge.

SECONDARY OUTCOMES:
Medical cost | at discharge 1 day, an average of 7days
  Direct medical cost at discharge
Radiation dose | during the procedure
  Amount of radiation dose
Time in the Cathlab | during the procedure
  Time in the Cathlab
Time for the TAVI procedure | during the procedure
  Time for the TAVI procedure
All-cause mortality and its sub-categories | at discharge 1 day, an average of 7days; 30-day; 1 year
  All-cause mortality and its sub-categories defined by VARC 3
All strokes | at discharge 1 day, an average of 7days;30-day; 1 year
  All strokes
Any hospitalization and its sub-categories | 30-day, 1 year
  Any hospitalization and its sub-categories defined by VARC 3
Acute Kidney Injury (AKI) | at discharge 1 day, an average of 7days; 30-day
  Acute Kidney Injury (AKI)(VARC 3 criteria: use the widely recognized kidney disease: Improving Global Outcomes (KDIGO) definition of AKI)
Type 3 (life-threatening) or Type 4 (leading to death) bleeding | at discharge 1 day, an average of 7days; 30-day; 1 year
  Type 3 (life-threatening) or Type 4 (leading to death) bleeding (VARC-3 criteria)
Mild or more prosthetic valve regurgitation | 30-day, 1 year
  Mild or more prosthetic valve regurgitation [TTE assessment
New permanent pacemaker implantation | at discharge 1 day, an average of 7days; 30-day, 1 year
  New permanent pacemaker implantation [VARC-3 criteria]
Conduction disturbances and arrhythmias | at discharge 1 day, an average of 7days; 30-day; 1 year
  Conduction disturbances and arrhythmias according to VARC-3
Technical success: | patient exit from procedure room,whichever came first,assessed up to 30 minutes
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the devicea or to a major vascular or access-related, or cardiac structural complication
Device success | 30-day
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the devicea or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valvec (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index >_0.25, and less than moderate aortic regurgitation)
Myocardial infarction | at discharge 1 day, an average of 7days; 30-day; 1 year
  Myocardial infarction (VARC-3 criteria)
Vascular and access-related complications | at discharge 1 day, an average of 7days; 30-day; 1 year
  Vascular and access-related complications (VARC-3 criteria)
Cardiac structural complications | at discharge 1 day, an average of 7days; 30-day; 1 year
  Cardiac structural complications (VARC-3 criteria)
Any adverse events | within 7 days
  Any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, PhD, Study Chair — Xijing Hospital, Xi'an, Shannxi, China; Junbo Ge, PhD, Principal Investigator — Zhongshan hospital, Fudan University, Shanghai, China; Patrick Washington Serruys, PhD, Study Chair — National University of Ireland Galway, Galway, Ireland; Yoshinobu Onuma, Ph D, Study Chair — National University of Ireland Galway, Galway, Ireland; Daxin Zhou, PhD, Study Chair — Zhongshan hospital, Fudan University, Shanghai, China; Rutao Wang, PhD, Study Chair — Xijing Hospital, Xi'an, Shannxi, China
Locations (2):
- China (2):
  - Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xijing hospital, Xi'an, Shannxi

IPD SHARING:
Plan to Share IPD: No